CLINICAL TRIAL: NCT05700578
Title: Evaluation of a Novel Behavior Change Intervention for Posttraumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Carter Bedford, Graduate Research Assistant, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002835
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: PTSD
Keywords: Psychoeducation; Online Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to complete one of two web based interventions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Elimination for Traumatic Stress (SBETS) (Experimental): Web-Based Safety Behavior Elimination for Traumatic Stress Intervention. (1) 30-minute session focused on providing psychoeducation about the nature of posttraumatic stress disorder (PTSD), how trauma-related safety behavior use worsens PTSD, and strategies to reduce or eliminate safety behavior use
  Interventions: Behavioral: Safety Behavior Elimination for Traumatic Stress (SBETS)
- Modifiable Behavior Intervention (MoBI) (Active Comparator): Web-Based Modifiable Behavior Intervention. (1) 30-minute session focused on providing psychoeducation about strategies to maintain one's physical and mental health, such as by exercising, maintaining a healthy diet, and managing stress.
  Interventions: Behavioral: Modifiable Behavior Intervention (MoBI)

INTERVENTIONS:
Behavioral: Safety Behavior Elimination for Traumatic Stress (SBETS) — This intervention took 30 minutes to complete. At the end of the intervention, participants were instructed to select two of their most commonly-used trauma-related safety behaviors to reduce or eliminate over the coming month.
  Arms: Safety Behavior Elimination for Traumatic Stress (SBETS)
Behavioral: Modifiable Behavior Intervention (MoBI) — The intervention took 30 minutes to complete. At the end of the intervention, participants were instructed to select two of their most commonly-used unhealthy behaviors to reduce or eliminate over the coming month.
  Arms: Modifiable Behavior Intervention (MoBI)

SUMMARY:
Evaluation of a Novel Behavior Change Intervention for Posttraumatic Stress

DETAILED DESCRIPTION:
This study compared exposure to one of two web-based treatments in self-reported improvement of posttraumatic stress disorder (PTSD) symptoms in adults with at least one lifetime traumatic event and elevated posttraumatic stress symptoms.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking individuals
* Experience of at least one lifetime traumatic event, as measured by the Life Events Checklist
* Score of 25 or higher on the PTSD Checklist for DSM-5

Exclusion Criteria:

* Pregnant women
* Adults unable to consent
* Prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to 2 weeks, change from baseline to 1 month
  A 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. 0-4 scale (0="Not at all", 1="A little bit", 2=" Moderately", 3="Quite a bit", and 4="Extremely.") A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.
Posttraumatic Safety Behavior Questionnaire (PSBQ) | Change from baseline to 2 weeks, change from baseline to 1 month
  A 23-item self-report measure assessing frequency of use of 23 trauma-related safety behaviors. 0-4 scale (0="Never", 1="Rarely", 2=" Sometimes", 3="Often", and 4="Always.") A total safety behavior use score (range - 0-92) can be obtained by summing the scores for each of the 23 items.

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Schmidt, Principal Investigator — Florida State University
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT05700578/ICF_000.pdf